CLINICAL TRIAL: NCT02779296
Title: Trial Investigating Cyanoacrylate Glue to Prevent Surgical Site Infection Following Breast Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OHSN-REB #20160009-01H
Record Dates: First submitted 2016-05-02; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Surgical Wound Infection
Keywords: Cyanoacrylates; Mammaplasty; Mastectomy
MeSH Terms: conditions — Surgical Wound Infection | interventions — octyl 2-cyanoacrylate; Tissue Adhesives

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2-Octyl Cyanoacrylate Glue (Experimental): At the surgical site, a thin layer of cyanoacrylate glue will be applied over the sutures at the time of closure.
  Interventions: Other: 2-Octyl Cyanoacrylate Glue
- No Glue (No Intervention): No cyanoacrylate glue will be applied.

INTERVENTIONS:
Other: 2-Octyl Cyanoacrylate Glue — topical
  Other Names: DERMABOND®; LIQUIBAND Exceed™; Tissue Adhesive; Dermal Glue
  Arms: 2-Octyl Cyanoacrylate Glue

SUMMARY:
Surgical Site Infections (SSI) represents a significant complication in plastic surgery. Infections can result in a prolonged recovery and impair long-term cosmetic appearance. One potential method to reduce infection is by applying a thin layer of dermal glue over the sutures at the site of incision immediately after the surgery. Conventional closures, such as sutures or staples, leave the site vulnerable until epithelialization occurs in 24 to 48 hours. In contrast, dermal glue provides an instant, waterproof barrier and it has been shown to have intrinsic bacteriostatic properties. The glue is supplied as a liquid enclosed in a vial and when applied, polymerizes rapidly in an exothermic reaction in the presence of moisture to form a solid adhesive. 2-Octylcyanoacrylate (2-OCA)-based glue is formulated to be more flexible than previous preparations. The application of dermal glue is rapid, simple and requires no specific follow-up as it naturally sloughs off overtime. The purpose of this study is to determine if 2-OCA-based glue can reduce the rate of surgical site infection following surgery. Patients undergoing breast surgery will be recruited and randomized to either a group receiving a layer of glue over sutures following surgery or no treatment. Patients will be followed up at 30 days and at 8 months for signs of infection, additional complications and the visual appearance of the scars. The cost of treating and infection will be calculated to determine if using dermal glue to prevent infection is economically feasible. This research has the potential to find a method to reduce surgical site infection, which can be applied to other surgeries.

ELIGIBILITY:
Inclusion Criteria:

* patient has provided signed consent
* undergoing surgery on the breast

Exclusion Criteria:

* Infection within 30 days
* Previous hypersensitivity to cyanoacrylates or formaldehyde

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 30 days post surgery

SECONDARY OUTCOMES:
Other Surgical Complications | 30 days post surgery
  Hematoma, seroma, wound dehiscence, scar hyperpigmentation, necrosis (nipple areolar complex, wound edges, fat tissue)
Other Surgical Complications | 8 months post surgery
  Hematoma, seroma, wound dehiscence, scar hyperpigmentation, necrosis (nipple areolar complex, wound edges, fat tissue)
Cosmetic Appearance assessed by the Patient and Observer Scar Assessment Scale (POSAS) v2.0 | 30 days post surgery
Cosmetic Appearance assessed by the Patient and Observer Scar Assessment Scale (POSAS) v2.0 | 8 months post surgery
Cost Analysis to determine the cost to treat a patient with and without a surgical site infection | 8 months post surgery
  This analysis will be conducted from a Ministry of Health perspective and will factor the additional cost of the glue with the additional cost of treating a surgical site infection (such as antibiotics, additional healthcare visits, treatments and procedures).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quinn JV, Osmond MH, Yurack JA, Moir PJ. N-2-butylcyanoacrylate: risk of bacterial contamination with an appraisal of its antimicrobial effects. J Emerg Med. 1995 Jul-Aug;13(4):581-5. doi: 10.1016/0736-4679(95)80025-5. PMID 7594385
- [Background] Hall LT, Bailes JE. Using Dermabond for wound closure in lumbar and cervical neurosurgical procedures. Neurosurgery. 2005 Jan;56(1 Suppl):147-50; discussion 147-50. doi: 10.1227/01.neu.0000144170.39436.52. PMID 15799803